CLINICAL TRIAL: NCT01648556
Title: Research of Predictive Factors to Immune Thrombopenic Purpura in Front of a Thrombopenia in Appearance Isolated in the Elderly
Brief Title: Research of Predictive Factors to Immune Thrombopenic Purpura
Acronym: PREDI-PTI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2011_843_0002
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Purpura Thrombopenic
Keywords: Purpura thrombopenic; Medullary cytogenetics; Myelodysplasic syndrome; bone marrow biopsy
MeSH Terms: conditions — Purpura, Thrombocytopenic | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patients with a thrombopenia isolated (Other): Patients of 60 years old and more presenting a thrombopenia isolated with a rate of platelet < 100 G/l Blood tests and bone marrow biopsy repeated
  Interventions: Other: Blood tests and bone marrow biopsy repeated

INTERVENTIONS:
Other: Blood tests and bone marrow biopsy repeated — Blood tests are realized for the dosage of the TPO, the dosage of the antiplatelet antibodies, to measure isotopic lifetime of platelet.
  The test in corticoids by the prednisone per os is realized too. The bone marrow biopsy is realized at the inclusion and during follow-ups if the haemogram is abnormal.
  Other Names: The test in corticoids by the prednisone per os

SUMMARY:
It is about a multicentric study prospective of more than patients' 60 years with a thrombopenia isolated of less than 100 G/L blood platelet without cause found to estimate so certain examinations realized in the diagnosis (medullary cytogenetics, dosage of the TPO, the Anti-platelet antibodies, isotopic lifetime of platelet) are in favour of the diagnosis of PTI.

DETAILED DESCRIPTION:
It is about a multicentric study prospective of more than patients' 60 years with a thrombopenia isolated of less than 100 G/L blood platelet without cause found to estimate so certain examinations realized in the diagnosis (medullary cytogenetics, dosage of the TPO, the Anti-platelet antibodies, isotopic lifetime of platelet) are in favour of the diagnosis of PTI.

The principal endpoint is to evaluate if the medullary cytogenetics is the predictive factor of the diagnosis of PTI in front of a thrombopenia isolated in elderly.

The secondary endpoints are :

* to identify at the time of the diagnosis, the factors and/or predictive markers correlated in the final diagnosis of PTI or SMD
* to study the respective frequency of the PTI and the SMD in front of a thrombopenia seemingly isolated of the subject of more than 60 years.

  200 patients will be included. 160 patients should be assessable at the end of study by considering the excluded patients, the dead and the lost sight.They will be followed every 4 months, during two years.

In every visit, will be realized a clinical examination, a blood film, a haemogram.

If the haemogram is abnormal, a bone marrow biopsy is realized. The patient who presents a myelodysplastic syndrome is excluded.

ELIGIBILITY:
Inclusion Criteria:

* Rate of platelet < 100 G/l for less than 12 months ,
* age = ou > 60 years,
* haemoglobin > ou = 12 g / dl at the woman, > ou = 13 g/dl at the man,
* polymorphonuclear neutrophil > ou = 1.7 G/l,
* monocytes < ou= 1 G/l,
* lymphocytes < ou = à 4 G/l,
* VGM < 100 fL, blood film normal,
* informed consent,
* expectation of life > 6 months

Exclusion Criteria:

* hepatomegaly,
* splenomegaly,
* hepatic abnormality,
* blood coagulation abnormality,
* antecedent of auto-immune disease,
* drug thrombopenia,
* HIV, VHB or VHC positive,
* antecedent of malicious tumor in the 5 years before inclusion

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
the result of cytogenetics medullary | two years after inclusion
  the primary endpoint corresponds to the occurence of the PTI after two years after inclusion.

SECONDARY OUTCOMES:
dosage of the TPO | EVERY 4 MONTHS (followed every four months during two years apres inclusion)
the result to the antibodies antiplatelet (positive or negative) for MAIPA | EVERY 4 MONTHS (followed every 4 months during two years after the inclusion)
The isotopic lifetime of platelet | EVERY 4 MONTHS (followed every four months during two years apres inclusion)
  < or > 3.5 days
The test in corticoids by the prednisone per os | EVERY 4 MONTHS (followed every 4 months during two years after the inclusion)
  1 mg / kg / day for 3 weeks The therapeutic test is considered as positive if a number of platelets is > 50 G/l with at least a doubling of the platelet rate before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre MD MAROLLEAU, phD, Principal Investigator — CHU AMIENS; mathilde HUNAULT BERGER, Ph D, Principal Investigator — University Hospital, Angers; NADINE MAGY BERTRAND, PH D, Principal Investigator — Centre Hospitalier Universitaire de Besancon; Olivier FAIN, PH D, Principal Investigator — HOPITAL JEAN VERDIER, BONDY; BRIGITTE PAN PETESCH, D, Principal Investigator — CHU BREST; MICHEL LEPORRIER, PH D, Principal Investigator — University Hospital, Caen; BERTRAND GODEAU, PH D, Principal Investigator — CHU CRETEIL; PHILIPPE BIERLING, PH D, Principal Investigator — EFS IVRY SUR SEINE; LOUIS TERRIOU, PH D, Principal Investigator — CHRU LILLE; JEAN MARC DURAND, PH D, Principal Investigator — LA CONCEPTION MARSEILLE
Locations (1):
- CHU Amiens, Amiens, France